CLINICAL TRIAL: NCT03039387
Title: The Effect of Transcranial Direct Current Stimulation (tDCS) on Cognitive Control and Emotion Regulation in Depressed Patients
Brief Title: Effects of tDCS on Cognitive Control and Emotion Regulation in Depressed Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 01EE1403D
Record Dates: First submitted 2016-10-28; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-08

CONDITIONS: Anodal Stimulation tDCS; Major Depression; Cognitive Control; Emotion Regulation
MeSH Terms: conditions — Depressive Disorder, Major; Emotional Regulation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anodal tDCS (Active Comparator): transcranial direct current stimulation of the left dlPFC with 1mA
  Interventions: Device: anodal transcranial direct current stimulation
- Sham stimulation (Placebo Comparator): Double blind sham stimulation (stimulation will be ramped down after 30 sec.)
  Interventions: Device: transcranial direct current stimulation (sham)

INTERVENTIONS:
Device: anodal transcranial direct current stimulation
  Other Names: anodal tDCS
  Arms: anodal tDCS
Device: transcranial direct current stimulation (sham) — for the placebo control condition, the transcranial direct current stimulation will only last for 30 seconds and will then be ramped down.
  Other Names: sham tDCS
  Arms: Sham stimulation

SUMMARY:
Deficient cognitive control (CC) and the use of dysfunctional emotion regulation strategies (ERS) are both central characteristics of major depression. Both are associated with reduced activity of the dorsolateral prefrontal cortex (dlPFC). Transcranial direct current stimulation (tDCS) is a safe, simple and effective non-invasive method to modulate the cortical excitability. The goal of this randomized, sham-controlled, double blind clinical trial is to examine the effect of transcranial direct current stimulation (tDCS) on the CC and ERS in depressed patients compared to healthy subjects. Overall, the study will include 44 participants (22 depressed Patients and 22 healthy subjects). Each participant will complete a CC task while receiving sham tDCS in one session and anodal tDCS in the other session (counterbalanced). Afterwards the ERS 'rumination' will be measured during a resting phase by means of a questionnaire and psychophysiological measures (heart rate variability). The investigators hypothesize (a) an amelioration of CC by anodal tDCS and (b) a reduced use of the dysfunctional emotion regulation strategy 'rumination' after anodal tDCS. Overall this experiment will provide new and reliable data for the development of new treatment methods.

DETAILED DESCRIPTION:
1. Working hypothesis: anodal transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex (dlPFC) can enhance healthy and impaired cognitive control (CC) and reduce the use of dysfunctional emotion regulation strategies.
2. Previous work of the investigators: The investigators previous work has provided decisive evidence for polarity-specific activity-dependent effects of tDCS to the left dlPFC on cognitive planning and control of emotional information processing in healthy subjects and patients with MD. Particularly, reduced prefrontal brain activity during a working memory task in patients with MD was found by using near infrared spectroscopy (NIRS). In addition, the investigators demonstrated that a single session, anodal, activity enhancing tDCS to the left dlPFC ameliorates deficient CC in patients with depression, whereas cathodal, activity reducing tDCS, induces a depression-like negativity bias in healthy subjects. Furthermore, the investigators showed that during anodal tDCS of the left dlPFC healthy subjects showed (a) better performance in a CC task (b) no increase in angry mood after the task compared to a control group and (c) that elevated angry mood was associated to a worse performance in the CC task.
3. Aims and workplan: to investigate the effects of anodal tDCS of the left dLPFC in healthy and depressed subjects the investigators will conduct a double-blind, randomized, sham-controlled, cross-over design. In two sessions each participant (22 depressed and 22 healthy subjects, N= 44) will complete a CC task while receiving anodal tDCS (1 mA) to the left dlPFC in one session and sham tDCS in the other session (counterbalanced). Afterwards the ERS 'rumination' will be measured during a resting phase by means of a questionnaire and psychophysiological measures.

ELIGIBILITY:
Inclusion Criteria for depressed patients

* diagnosed major depression (DSM-V)
* stable medication for four weeks

Inclusion Criteria for all participants

* right handedness

Exclusion Criteria:

* history of seizures
* metal device throughout the body
* pregnancy
* use of von antipsychotics / mood stabilizer
* diagnosed bipolar disorder
* current substance abuse (nicotine excluded)
* diagnosed psychotic diseases
* diagnosed anorexia nervosa
* diagnosed personality disorders: cluster A, antisocial personality disorder, borderline personality disorder

Exclusion Criteria for healthy participants:

* history of affective disorders or current affective disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Interstimulusintervall and number of correct trials in the PASAT | Assessment during stimulation/ sham stimulation in two sessions through study completion, on average 10 days.
  To measure the performance in the PASAT the number of correct trials as well as the mean Interstimulusintervall will be assessed.
Change of positive and negative affect | The positive and negative affect is assessed (a) right before and after the PASAT in two sessions through study completion, on average 10 days. And (b) also after the resting phase in two sessions through study completion, on average 10 days.
  Change of positive and negative affect after, compared to before performing the PASAT and also change of the affect during the resting phase.
Heart rate variability | in two sessions through study completion, on average 10 days
  The Heart Rate Variability will be measured during the resting phase right after the measurement of the affect.
Score in state rumination questionnaire | in two sessions through study completion, on average 10 days
  The state rumination will be measured after the resting phase

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No